CLINICAL TRIAL: NCT03754088
Title: Initiation of an in Vitro Model of the Cystic Fibrosis Bronchial Epithelium Via Induced Pluripotent Stem Cell Technology
Brief Title: In Vitro Model of the Cystic Fibrosis Bronchial Epithelium Via iPS Technology
Acronym: PaCyFIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0254; 2017-A02341-52 (Other: RCB number)
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2021-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, RNA and induced pluripotent stem cell lines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis: Three cystic fibrosis patients who are homozygous for the p.Phe508del mutation.
- Healthy subjects: Three healthy subjects.

SUMMARY:
In order to further enable physiopathology studies, the aim of this project is to validate an in vitro model of cystic fibrosis created using induced pluripotent stemcell (iPS) differentiated bronchial epithelium from cystic fibrosis (CF) patients homozygous for the p.Phe508del mutation of the cystic fibrosis transmembrane conductance regulator (CFTR) gene.

DETAILED DESCRIPTION:
The investigator's primary objective is to generate iPS lines from 3 CF patients and from 3 healthy subjects.

Secondary objectives include verification that cell lines express the CFTR gene according to their genotype, verification or relative production of the CFTR protein for each iPS line, and amplification of obtain iPS lines for aliquot creation to facilitate sharing.

ELIGIBILITY:
Inclusion Criteria for subjects with Cystic Fibrosis:

* Homozygote for the p.Phe508del mutation
* Signed informed consent given by the subject

Inclusion Criteria for subjects without Cystic Fibrosis:

* Signed informed consent given by the subject

Exclusion Criteria:

* Pregnancy, breastfeeding
* Participant in an exclusion period determined by a previous study
* Participant under any kind of guardianship
* Unaffiliated with or not a beneficiary of a social security program (health insurance)
* Subject deprived of liberty (e.g. prisoners)
* Subject with positive infectious markers for HIV1, HIV2, HBC or HBV

Exclusion Criteria for subjects with Cystic Fibrosis:

* Any pathology requiring a treatment or a pathology not requiring treatment but with clinical significance according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three cystic fibrosis patients who are homozygous for the p.Phe508del mutation and 3 healthy subjects without cystic fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Obtention of induced pluripotent stem cell line (iPS): yes/no | 28 days
  Was a pluripotent stem cell line obtained? yes/no

SECONDARY OUTCOMES:
Functional bronchial epithelium present for the iPS? yes/no | 28 days
  Was a functional bronchial epithelium present for the iPS? yes/no
Cystic fibrosis transmembrane conductance regulator (CFTR) channel function: yes/no | 28 days
  CFTR channel function demonstrated via response following exposure to modified oligonucleotides targeting the mutated CFTR transcript.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD, PhD, Principal Investigator — Montpellier University Hospitals
Locations (1):
- Hôpital Arnaud de Villeneuve - CHU de Montpellier, Montpellier, France